CLINICAL TRIAL: NCT02368171
Title: Role of Heme-oxygenase (HO) and Nitric Oxide (NO) Pathway in Patients With Obstructive Sleep Apnea (OSA) and Pulmonary Hypertension (PH)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Behrouz Jafari, Assisstant professore of medicine, Southern California Institute for Research and Education
Other Study IDs: OSA-PH-001
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Obstructive Sleep Apnea; Pulmonary Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension, Pulmonary | interventions — Nitric Oxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Obstructive sleep apnea with pulmonary hypertension: Patients with AHI> 5/h and pulmonary hypertension with RVSP>35 mmHg on Echo
  Interventions: Other: measure exhaled carbon monoxide and nitric oxide
- control: patients with AHI<5/h and RVSP<35 mmHg on Echo
  Interventions: Other: measure exhaled carbon monoxide and nitric oxide
- OSA with no Pulmonary hypertension: patients with AHI>5/h, but RVSP<35 mmHg on Echo
  Interventions: Other: measure exhaled carbon monoxide and nitric oxide

INTERVENTIONS:
Other: measure exhaled carbon monoxide and nitric oxide

SUMMARY:
Research design: This is a controled prospective study.

Methodology:

Patients with newly diagnosed and untreated OSA with total apnea-hypopnea index (AHI) >5/h, and control (AHI<5/h) will be recruited from the Long Beach VA sleep center. Controls are subjects without OSA or other sleep disorders and no sign of pulmonary hypertension based on echo. The investigators also measure pulmonary artery pressure by 2D Echo and exclude patient with any sign of left heart dysfunction. PH will be defined as RVSP > 35 mmHg or mean PA pressure>25 mmHg. The investigators will recruit subjects with and without PH and OSA in three separate groups:

1. group one : OSA+ PH,
2. group two: normal individual with no OSA and no PH,
3. group three: OSA with no PH Pulmonary function test will be done to exclude patients with underlying lung disease.

The inclusion criteria is: Age >20, AHI >5, AHI <5 (as control), RVSP > 35 mmHg OR Mean PA pressure>25 mmHg, RVSP < 35 mmHg OR Mean PA pressure < 25 mmHg (as control).

Subjects will be excluded if they had known peripheral vascular disease, liver disease, hemolytic anemia, inflammatory disease, active infection, or if they were pregnant, on therapy for OSA, on chronic steroid treatment, or younger than 20 years of age, patients with left heart failure (systolic or diastolic), patients are on PH medications including sildenafil, active smokers, COPD and asthma, active infection or inflammatory disease and collagen vascular disease.

Nocturnal polysomnography will be performed and scored according to the American Academy of Sleep Medicine.

Exhaled Carbon monoxide (CO) will be measured with a calibrated fuel cell type electrochemical device with sensor sensitivity of 1 ppm. The mean of three reproducible measurements will be recorded and corrected for ambient CO.

Exhaled Nitric Oxide (NO) will be measured. At each testing session, at least three flow-regulated FENO measurements will be performed.

The investigators will repeat 2D Echo and measurements of above factors after 3 months of CPAP treatment. The investigators also check patient's compliance with the treatment by downloading data off of their CPAP device.

Each subject will be informed of the experimental procedures, which is approved by the Human Investigation Committee of the VA-Long Beach.

Finding:

The investigators hypothesize that HO pathway causing perturbation of pulmonary endothelial function by inhibition of nitric oxide.

Clinical significance:

OSA is associated with PH, but exact mechanism is not well known. In the past, I have shown that increased endogenous CO in the setting of elevated NO concentration is associated with endothelial dysfunction in patient with OSA. Therefore, the investigators sought to investigate the roles of HO and NO pathways in patients with OSA associated with PH.

Impact/significance:

It addresses a fundamental gap in our understanding of how OSA results in increase the pulmonary artery pressure and if substantiated, will provide the basis for the design and testing of new approaches to prevention and treatment of OSA.

ELIGIBILITY:
Inclusion Criteria:

1. participants must satisfy diagnostic criteria for Obstructive sleep apnea.
2. evidence of pulmonary hypertension disease base upon one or more of the following: RVSP > 35 mmHg OR Mean PA pressure>25 mmHg, RVSP < 35 mmHg OR Mean PA pressure < 25 mmHg (as control).
3. age greater than or equal to 20 years.
4. no significant alcohol use (7 or fewer drinks per week).

Exclusion Criteria:

1. peripheral vascular disease
2. liver disease
3. Pregnancy. A serum pregnancy test must be performed and negative in all women of child bearing potential within 2 weeks prior to enrollment.
4. Any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation, and compliance with the study criteria.
5. hemolytic anemia
6. inflammatory disease
7. active infection,
8. on therapy for OSA,
9. on chronic steroid treatment,
10. younger than 20 years of age,
11. patients with left heart failure (systolic or diastolic),
12. patients are on pulmonary hypertension medications including sildenafil,
13. active smokers,
14. COPD and asthma,
15. active infection or inflammatory disease
16. collagen vascular disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed and untreated OSA with total apnea-hypopnea index (AHI) >5/h, and control (AHI<5/h) will be recruited from the Long Beach VA sleep center. Controls are subjects without OSA or other sleep disorders and no sign of pulmonary hypertension based on echo. We also measure pulmonary artery pressure by 2D Echo and exclude patient with any sign of left heart dysfunction. PH will be defined as RVSP > 35 mmHg or mean PA pressure>25 mmHg. We will recruit subjects with and without PH and OSA in three separate groups:
  1. group one : OSA+ PH,
  2. group two: normal individual with no OSA and no PH,
  3. group three: OSA with no PH Pulmonary function test will be done to exclude patients with underlying lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
exhaled carbon monxide and nitric oxide | 3 month
  The concentration of both gas will be measured in PPM and will be repeated in 3 month after CPAP is being used.
RVSP as sorrogate of Pulmonary artery pressure | 3 month
  It will be measured by 2D-Echo in mmHg and correlation of RVSP and above two gases will be assessed.